CLINICAL TRIAL: NCT03499821
Title: A Multicenter Clinical Evaluation of the Clinical Performance of a Phakic Intraocular Lens
Brief Title: Clinical Performance of a Phakic Intraocular Lens (IOL)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Staar Surgical Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Study CP17-01
Record Dates: First submitted 2018-04-09; First posted 2018-04-17 (Actual); Results first posted 2022-09-21 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Intervention Model Description: Device: Open label, all subjects receive same treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Study population (Experimental): EDOF ICL implanted into both eyes of eligible subjects.
  Interventions: Device: EDOF ICL

INTERVENTIONS:
Device: EDOF ICL — The Visian ICL is intended to be implanted within the posterior chamber, directly behind the iris, and in front of the anterior capsule of the human crystalline lens. It offers an intraocular alternative for the correction of refractive error in those who currently utilize spectacle and/or contact lenses correction.
  Other Names: EVO+ Visian ICL with Aspheric (EDOF) Optic

SUMMARY:
This study will evaluate the clinical performance of a phakic intraocular lens (IOL) for the improvement of Uncorrected Near Visual Acuity (UCNVA) in subjects who require between +1.00 and +2.50 Reading Add.

DETAILED DESCRIPTION:
This is a prospective, open-labeled, multi-site evaluation of clinical performance of the STAAR EVO+ Visian™ Implantable Collamer® Lens (VICL) with Aspheric (EDOF) Optic [EDOF ICL] for the improvement of UCNVA in subjects who require between +1.00 and +2.50 Reading Add.

Approximately 48 subjects who meet all eligibility criteria will undergo EDOF ICL implantation in both eyes. All eyes will be followed for 6 months after surgery.

The first eye implanted with the study lens and the appropriate time for fellow eye implantation will be determined by the medical judgement of the Investigator. All eyes will be analyzed for safety and performance.

The primary performance endpoint is defined as achievement of monocular UCNVA of Snellen equivalent 20/40 or better at 40 cm at 6 months after implantation in equal to or greater than 75% of implanted eyes.

ELIGIBILITY:
Inclusion Criteria:

1. Must be able to read, understand and provide written informed consent,
2. Willing and able to comply with all treatment and follow-up study related procedures,
3. 40 - 60 years of age at time of surgery if require spherical lens powers from -0.50 D to -18.00 D,
4. 35 - 45 years of age at time of surgery if require a spherical lens power from 0.0 D to +3.00 D,
5. Preoperative refraction fully correctable with available lens powers, with ≤ 0.75 D preoperative refractive and residual cylinder,
6. < 0.75 D spherical equivalent difference between cycloplegic and manifest refractions,
7. Stable correction (± 0.50 D) as determined by manifest refraction spherical equivalent (MRSE),
8. Best Corrected Distance Visual Acuity 20/20 or better in both eyes,
9. Requires +1.00 D to +2.50 D reading add,
10. Anterior chamber depth (ACD) ≥ 2.8 mm if require spherical lens powers from -0.50 D to -18.00 D,
11. ACD ≥ 3.0 mm if require spherical lens powers from 0.00 D to +3.00 D,
12. Anterior chamber angle ≥ Grade III,
13. Phakic in both eyes,
14. Current contact lens wearers need to demonstrate a stable refraction, (± 0.5 D), expressed as MRSE, on two consecutive examination dates with refractive stability determined by the following criteria:

    1. contact lenses were not worn for at least 2 weeks (rigid and toric contact lenses) or 3 days (soft contact lenses) prior to the first refraction,
    2. two refractions were performed at least 7 days apart.

Exclusion Criteria:

1. Participation in a clinical trial within 30 days prior to entry into this study and/or during the period of study participation,
2. Previous intraocular or corneal surgery in either eye, including refractive surgery,
3. Progressive sight threatening disease or other previous or current ocular conditions, other than myopia in either eye,
4. Low/abnormal corneal endothelial cell density,
5. Amblyopia,
6. Presence of active or history of chronic inflammation in either eye,
7. Clinically significant irregular astigmatism in either eye,
8. Serious, acute, chronic or systemic, non-ophthalmic disease or illness that would increase the operative risk, confound the outcome(s) of the study or which may preclude study completion,
9. Use of topical steroids at time of implantation,
10. Systemic or topical medication, other than prescribed study medications that may confound the outcome or increase the risk to the subject,
11. Allergy to anesthetics or other postoperative medications required in this study,
12. Subject who is pregnant, plans to become pregnant, or is lactating during the course of the study, or has another condition associated with the fluctuation of hormones that could lead to refractive changes,
13. Subjects who present any emotional, physiologic, or anatomical condition which may preclude study participation.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2019-07-09 (Actual); Study Completion 2019-07-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Egamino, PhD, Study Director — Staar Surgical Company
Locations (6):
- Mediopolis, Antwerp, Belgium
- Spain (5):
  - Instituto Oftalmológico Fernández-Vega, Oviedo, Principality of Asturias
  - Qvision-Hospital Vithas Virgen del Mar, Almería
  - IMO Instituto de Microcirugía Ocular, Barcelona
  - Innova Ocular Begitek, San Sebastián
  - Clínica Oftalmológica Gasteiz, Vitoria-Gasteiz

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Packer M, Alfonso JF, Aramberri J, Elies D, Fernandez J, Mertens E. Performance and Safety of the Extended Depth of Focus Implantable Collamer(R) Lens (EDOF ICL) in Phakic Subjects with Presbyopia. Clin Ophthalmol. 2020 Sep 18;14:2717-2730. doi: 10.2147/OPTH.S271858. eCollection 2020. PMID 32982164

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 41 subjects were screened in the study. Six did not meet eligibility and 35 subjects were treated at 6 clinical sites in Europe (5 sites in Spain and 1 site in Belgium). The first enrolled subject underwent bilateral surgery in May 2018, the last subject completed the last study visit in July 2019.
Units Other Than Participants: eyes
Groups:
- Study Population: Extended Depth of Field (EDOF) Implantable Collamer Lens (ICL) implanted into both eyes of eligible subjects.
  EDOF ICL: The Visian ICL is intended to be implanted within the posterior chamber, directly behind the iris, and in front of the anterior capsule of the human crystalline lens. It offers an intraocular alternative for the correction of refractive error in those who currently utilize spectacle and/or contact lenses correction.
Period: Overall Study
Arm/Group | Study Population
Started | 35; 70 eyes
Completed | 34; 68 eyes
Not Completed | 1; 2 eyes

BASELINE CHARACTERISTICS:
Units Other Than Participants: eyes
Arm/Group | Study Population
Number analyzed (Participants) | 35
Number analyzed (eyes) | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 35
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 35
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 10
  Spain | 25
Monocular UNVA better than 20/40 at Preoperative Visit [Number; unit: Eyes] — Monocular uncorrected near visual acuity (UNVA) at Preoperative Visit
  Eyes | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Eyes With Monocular Uncorrected Near Visual Acuity of 20/40 or Better at 40 cm 6 Months After Implantation
Description: Number of Eyes with Monocular Uncorrected Near Visual Acuity of 20/40 or better at 40 cm six months after implantation
Time Frame: 6 months
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Study Population
Number analyzed (Participants) | 34
Number analyzed (Eyes) | 68
Eyes | 66

2. Secondary Outcome: Percentage of Implanted Eyes Achieving Monocular Uncorrected Near Visual Acuity of 20/40 or Better at 40 cm 1 Month After Implantation
Description: Percentage of implanted eyes achieving Monocular Uncorrected Near Visual Acuity (UNVA) of 20/40 or better at 40 cm 1 month after implantation
Time Frame: 1 month
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Study Population
Number analyzed (Participants) | 34
Number analyzed (Eyes) | 68
Eyes | 66

3. Secondary Outcome: Percentage of Implanted Eyes Achieving Monocular Uncorrected Near Visual Acuity of 20/40 or Better at 40 cm 3 Months After Implantation
Description: Percentage of implanted eyes achieving Monocular Uncorrected Near Visual Acuity (UNVA) of 20/40 or better at 40 cm 3 months after implantation
Time Frame: 3 months
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Study Population
Number analyzed (Participants) | 34
Number analyzed (Eyes) | 68
Eyes | 66

4. Secondary Outcome: Change From Baseline in Monocular Uncorrected Intermediate Visual Acuity at 80 cm 1 Month Post Implantation
Description: Change from baseline in Monocular Uncorrected Intermediate Visual Acuity (UIVA) at 80 cm 1 month post implantation
Time Frame: Baseline and 1 month
Measure: Mean (Standard Deviation); unit: Lines of Vision Gained
Units Other Than Participants: Eyes
Arm/Group | Study Population
Number analyzed (Participants) | 34
Number analyzed (Eyes) | 68
Lines of Vision Gained | 7.63 (3.42)

5. Secondary Outcome: Change From Baseline in Monocular Uncorrected Intermediate Visual Acuity at 80 cm 3 Months Post Implantation
Description: Change from baseline in Monocular Uncorrected Intermediate Visual Acuity (UIVA) at 80 cm 3 months post implantation
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: Lines of Vision Gained
Units Other Than Participants: Eyes
Arm/Group | Study Population
Number analyzed (Participants) | 34
Number analyzed (Eyes) | 68
Lines of Vision Gained | 7.69 (3.48)

6. Secondary Outcome: Change From Baseline in Monocular Uncorrected Intermediate Visual Acuity at 80 cm 6 Months Post Implantation
Description: Change from baseline in Monocular Uncorrected Intermediate Visual Acuity (UIVA) at 80 cm 6 months post implantation
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: Lines of Vision Gained
Units Other Than Participants: Eyes
Arm/Group | Study Population
Number analyzed (Participants) | 34
Number analyzed (Eyes) | 68
Lines of Vision Gained | 7.79 (3.53)

7. Secondary Outcome: Change From Baseline in Monocular Uncorrected Near Visual Acuity at 40 cm 1 Month Post Implantation
Description: Change from baseline in Monocular Uncorrected Near Visual Acuity (UNVA) at 40 cm 1 month post implantation
Time Frame: Baseline and 1 month
Measure: Mean (Standard Deviation); unit: Lines of Vision Gained
Units Other Than Participants: Eyes
Arm/Group | Study Population
Number analyzed (Participants) | 34
Number analyzed (Eyes) | 68
Lines of Vision Gained | 5.96 (3.9)

8. Secondary Outcome: Change From Baseline in Monocular Uncorrected Near Visual Acuity at 40 cm 3 Months Post Implantation
Description: Change from baseline in Monocular Uncorrected Near Visual Acuity (UNVA) at 40 cm 3 months post implantation
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: Lines of Vision Gained
Units Other Than Participants: Eyes
Arm/Group | Study Population
Number analyzed (Participants) | 34
Number analyzed (Eyes) | 68
Lines of Vision Gained | 5.93 (4.05)

9. Secondary Outcome: Change From Baseline in Monocular Uncorrected Near Visual Acuity at 40 cm 6 Months Post Implantation
Description: Change from baseline in Monocular Uncorrected Near Visual Acuity (UNVA) at 40 cm 6 months post implantation
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: Lines of Vision Gained
Units Other Than Participants: Eyes
Arm/Group | Study Population
Number analyzed (Participants) | 34
Number analyzed (Eyes) | 68
Lines of Vision Gained | 6.22 (3.95)

10. Secondary Outcome: Change From Baseline in Monocular Distance Corrected Intermediate Visual Acuity at 80 cm 1 Month Post Implantation
Description: Change from baseline in Monocular Distance Corrected Intermediate Visual Acuity (DCIVA) at 80 cm 1 month post implantation
Time Frame: Baseline and 1 month
Measure: Mean (Standard Deviation); unit: Lines of Vision Gained
Units Other Than Participants: Eyes
Arm/Group | Study Population
Number analyzed (Participants) | 34
Number analyzed (Eyes) | 68
Lines of Vision Gained | .24 (2)

11. Secondary Outcome: Change From Baseline in Monocular Distance Corrected Intermediate Visual Acuity at 80 cm 3 Months Post Implantation
Description: Change from baseline in Monocular Distance Corrected Intermediate Visual Acuity (DCIVA) at 80 cm 3 months post implantation
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: Lines of Vision Gained
Units Other Than Participants: Eyes
Arm/Group | Study Population
Number analyzed (Participants) | 34
Number analyzed (Eyes) | 68
Lines of Vision Gained | .31 (2.02)

12. Secondary Outcome: Change From Baseline in Monocular Distance Corrected Intermediate Visual Acuity at 80 cm 6 Months Post Implantation
Description: Change from baseline in Monocular Distance corrected intermediate visual acuity (DCIVA) at 80 cm 6 months post implantation
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: Lines of Vision Gained
Units Other Than Participants: Eyes
Arm/Group | Study Population
Number analyzed (Participants) | 34
Number analyzed (Eyes) | 68
Lines of Vision Gained | .44 (2.09)

13. Secondary Outcome: Change From Baseline in Monocular Distance Corrected Near Visual Acuity at 40 cm 1 Month Post Implantation
Description: Change from baseline in Monocular Distance Corrected Near Visual Acuity (DCNVA) at 40 cm 1 month post implantation
Time Frame: Baseline and 1 month
Measure: Mean (Standard Deviation); unit: Lines of Vision Gained
Units Other Than Participants: Eyes
Arm/Group | Study Population
Number analyzed (Participants) | 34
Number analyzed (Eyes) | 68
Lines of Vision Gained | 1 (1.6)

14. Secondary Outcome: Change From Baseline in Monocular Distance Corrected Near Visual Acuity at 40 cm 3 Months Post Implantation
Description: Change from baseline in Monocular Distance Corrected Near Visual Acuity (DCNVA) at 40 cm 3 months post implantation
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: Lines of Vision Gained
Units Other Than Participants: Eyes
Arm/Group | Study Population
Number analyzed (Participants) | 34
Number analyzed (Eyes) | 68
Lines of Vision Gained | .92 (1.74)

15. Secondary Outcome: Change From Baseline in Monocular Distance Corrected Near Visual Acuity at 40 cm 6 Months Post Implantation
Description: Change from baseline in Monocular Distance Corrected Near Visual Acuity (DCNVA) at 40 cm 6 months post implantation
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: Lines of Vision Gained
Units Other Than Participants: Eyes
Arm/Group | Study Population
Number analyzed (Participants) | 34
Number analyzed (Eyes) | 68
Lines of Vision Gained | 1.11 (1.62)

16. Secondary Outcome: Change From Baseline in Binocular Uncorrected Near Visual Acuity at 40 cm 1 Month Post Implantation
Description: Change from baseline in Binocular Uncorrected Near Visual Acuity (UNVA) at 40 cm 1 month post implantation
Time Frame: Baseline and 1 month
Measure: Mean (Standard Deviation); unit: Lines of Vision Gained
Arm/Group | Study Population
Number analyzed (Participants) | 34
Lines of Vision Gained | 5.95 (3.99)

17. Secondary Outcome: Change From Baseline in Binocular Uncorrected Near Visual Acuity at 40 cm 3 Months Post Implantation
Description: Change from baseline in Binocular Uncorrected Near Visual Acuity (UNVA) at 40 cm 3 months post implantation
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: Lines of Vision Gained
Arm/Group | Study Population
Number analyzed (Participants) | 34
Lines of Vision Gained | 5.99 (4.01)

18. Secondary Outcome: Change From Baseline in Binocular Uncorrected Near Visual Acuity at 40 cm 6 Months Post Implantation
Description: Change from baseline in Binocular Uncorrected Near Visual Acuity (UCNVA) at 40 cm 6 months post implantation
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: Lines of Vision Gained
Arm/Group | Study Population
Number analyzed (Participants) | 34
Lines of Vision Gained | 6.12 (3.96)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Study Population
All-Cause Mortality (participants affected / at risk) | 0/35
Serious Adverse Events (participants affected / at risk) | 9/35
Other Adverse Events (participants affected / at risk) | 13/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Population (N=35)
Visual Acuity Reduced (Eye disorders) | 9 (11)
Vascular Migraine with Aura (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Population (N=35)
Visual Acuity Reduced (Eye disorders) | 8 (12)
Dry Eye (Eye disorders) | 5 (5)
Corneal Oedema (Eye disorders) | 2 (2)
Eye Pruritus (Eye disorders) | 1 (1)
Eye Inflammation (Eye disorders) | 1 (1)
Lacrimation Increased (Eye disorders) | 1 (1)
Hordeolum (Infections and infestations) | 2 (4)
Conjunctivitis (Infections and infestations) | 1 (1)
Intraocular Pressure Increased (Investigations) | 3 (3)
Conjunctival Laceration (Injury, poisoning and procedural complications) | 1 (1)

LIMITATIONS AND CAVEATS:
The study included subjects with residual accommodation. In order to further elucidate the performance of the EDOF ICL vis a vis severity of presbyopia at baseline, the performance of those eyes and subjects which not only required a reading add but also exhibited distance corrected near visual acuity of 20/40 or worse at baseline was examined. Refer to publication in reference module for more details.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data generated from the study will be regarded as confidential, until appropriate analysis and review by the Sponsor or its designee are completed. The results of the study may be published or presented by the Investigator(s) after review by, and in consultation and agreement with the Sponsor, and such that confidential or proprietary information is not disclosed. Prior to publication or presentation, a copy of the final text should be forwarded to the Sponsor or designee for comment.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-14): https://cdn.clinicaltrials.gov/large-docs/21/NCT03499821/Prot_SAP_000.pdf